CLINICAL TRIAL: NCT00158782
Title: An Open-Label, Safety, Pharmacokinetic and Pharmacodynamic Study of Multiple Doses of GW786034 and Lapatinib Concomitantly Administered in Cancer Patients
Brief Title: Study Of Safety And Tolerability Of GW786034 Given With Lapatinib In Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEG10006
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Carcinoma, Renal Cell
Keywords: Cancer GW786034 Lapatinib Pazopanib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Cohort 1 (Experimental): Subjects will receive GW786034 500 milligrams and lapatinib 750 milligrams.
  Interventions: Drug: GW786034; Drug: lapatinib
- Cohort 2 (Experimental): Subjects will receive GW786034 250 milligrams and lapatinib 750 milligrams.
  Interventions: Drug: GW786034; Drug: lapatinib
- Cohort 3 (Experimental): Subjects will receive GW786034 250 milligrams and lapatinib 1000 milligrams.
  Interventions: Drug: GW786034; Drug: lapatinib
- Cohort 4 (Experimental): Subjects will receive GW786034 500 milligrams and lapatinib 1000 milligrams.
  Interventions: Drug: GW786034; Drug: lapatinib
- Cohort 5 (Experimental): Subjects will receive GW786034 250 milligrams and lapatinib 1250 milligrams.
  Interventions: Drug: GW786034; Drug: lapatinib
- Cohort 6 (Experimental): Subjects will receive GW786034 400 milligrams and lapatinib 1250 milligrams.
  Interventions: Drug: GW786034; Drug: lapatinib
- Cohort 7 (Experimental): Subjects will receive GW786034 200 milligrams and lapatinib 1500 milligrams.
  Interventions: Drug: GW786034; Drug: lapatinib
- Cohort 8 (Experimental): Subjects will receive GW786034 400 milligrams and lapatinib 1500 milligrams.
  Interventions: Drug: GW786034; Drug: lapatinib
- Cohort 9 (Experimental): Subjects will receive GW786034 400 milligrams and lapatinib 1000 milligrams.
  Interventions: Drug: GW786034; Drug: lapatinib
- Cohort 10 (Experimental): Subjects will receive GW786034 800 milligrams and lapatinib 1500 milligrams.
  Interventions: Drug: GW786034; Drug: lapatinib

INTERVENTIONS:
Drug: GW786034 — GW786034 (Pazopanib) is an orally active, potent, reversible, small molecule tyrosine kinase inhibitor of vascular endothelial growth factor receptor 1 (VEGFR-1), VEGFR-2, VEGFR-3, platelet-derived growth factor receptor-alpha (PDGFR-alpha), PDGFR-beta, and c-Kit.
Drug: lapatinib — Lapatinib is an oral, reversible, tyrosine kinase inhibitor of both epidermal growth factor receptor-1 (ErbB1) and ErbB2.

SUMMARY:
This Phase I, dose finding study evaluates the safety and tolerability of lapatinib, a dual tyrosine kinase inhibitor, and GW786034, an anti-angiogenesis agent, when given together. The study first will find the best doses using safety and blood concentration data of both agents. This is done enrolling stepwise, cohorts of 3 patients each and the last patient enrolled must reach at least Day 22 of continuous daily dosing before the next cohort at an increased dose can begin. If a patient in a cohort has a dose limiting toxicity before Day 22, then 3 more patients are studied at that same dose. If 2 of 6 patients have dose limiting toxicities within the first 22 days, the next cohort receives the next lowest dose. Otherwise each cohort has an increasing dose of one of the two agents. The second stage of the study will administer the best doses of the agents to about 16 patients to further study safety and collect more blood concentration data (more blood samples in the second phase compared to the first phase). The second stage has the advantage of using the best dose (decreases chance of receiving a sub-therapeutic dose) while it collects more blood samples and requires slightly more long clinic visits.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed diagnosis of advanced solid tumor refractory to standard therapy or for whom there is no standard therapy.
* Females are eligible if they are of:

  a) Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who:
* had a hysterectomy.
* had a bilateral oophorectomy (ovariectomy).
* had a bilateral tubal ligation.
* is post-menopausal (a demonstration of total cessation of menses for 1 year).
* childbearing potential, has a negative serum pregnancy test at screening, and agrees to one of the following:
* an IUD with a documented failure rate of less than 1% per year.
* vasectomized partner who is sterile prior to the female patient's entry and is the sole sexual partner for that female.
* complete abstinence from sexual intercourse for 14 days before exposure to investigational product, throughout the clinical trial, and for at least 14 days after the last dose of investigational product.
* double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide).
* ECOG (Eastern Cooperative Oncology Group) PS 0 or 1.
* Adequate bone marrow function.
* Platelets greater than or equal to 75,000/mm3.
* ANC greater than or equal to 1,500/mm3 (1.5 x 109/L).
* Hgb greater than or equal to 9 g/dL (5 mmol/L).
* CLcr > 50 mL/min as calculated by the Cockcroft-Gault formula.
* Total bilirubin less than or equal to 1.5 x upper limit of normal.
* PT/INR/PTT less than or equal to 1.2 x upper limit of normal.
* AST/ALT less than or equal to 3 x upper limit of normal.
* Has LVEF within normal range or above 50% based on MUGA/ECHO.
* Urinalysis for protein is < 2 (negative, trace, or 1). NOTE: If urinalysis is 2 or greater then a 24 hour urine for protein must demonstrate less than 1 gram of protein in 24 hours for patient to be eligible for enrollment.
* Able to swallow and retain oral medication.
* Has a life expectancy of at least 12 weeks.

Exclusion criteria:

* Had prior treatment with either study drug.
* Has brain metastases.
* Uncontrolled hypertension (BP higher than 150/90 SBP/DBP).
* Have heart failure.
* Have DVT (deep vein thrombosis) or arterial thrombosis, MI (myocardial infarction), angina, or has had angioplasty and/or stenting within last 3 months.
* Has allergy to drug similar to lapatinib (e.g. allergic to Iressa(gefitinib) or Tarceva(erlotinib).
* Is using therapeutic doses of anti-coagulant.
* Has had major surgery, hormonal therapy, chemotherapy, radiotherapy, or other investigational agent within last 28 days.
* Pregnant or lactating.
* History or current GI (gastrointestinal) condition that alters stomach or gut emptying from normal (e.g. major surgery on the stomach).
* Bowel obstruction or chronic diarrhea.
* Psychological or geographical conditions that would prevent him/her from being a good candidate.
* Do not have accessible veins for venipuncture.
* History of prolonged QTc on ECG.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-09-28 (Actual); Primary Completion 2007-08-21 (Actual); Study Completion 2007-08-21 (Actual)

PRIMARY OUTCOMES:
Changes in pre and post treatment lab values and monitoring/reporting AES.AE's throughout study | throughout study
Labs every wk first cycle:day 1 subsequent cycles | first cycle:day 1 subsequent cycles

SECONDARY OUTCOMES:
find max conc of drugs in blood and time it occurs find out if drugs are taken up by the body, how much/for how long find out if drugs affect the size of the tumor. Blood taken day 15, 22 or 37 and tumor assessed every 8 wks | Blood taken day 15, 22 or 37 and tumor assessed every 8 wks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Durham, North Carolina, United States
- GSK Investigational Site, Rotterdam, Netherlands

REFERENCES:
- [Background] de Jonge MJ, Hamberg P, Verweij J, Savage S, Suttle AB, Hodge J, Arumugham T, Pandite LN, Hurwitz HI. Phase I and pharmacokinetic study of pazopanib and lapatinib combination therapy in patients with advanced solid tumors. Invest New Drugs. 2013 Jun;31(3):751-9. doi: 10.1007/s10637-012-9885-8. Epub 2012 Oct 6. PMID 23054212
- See also: Results for study VEG10006 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/VEG10006?search=study&study_ids=VEG10006#rs